CLINICAL TRIAL: NCT05024864
Title: HELicobacter Pylori Screening to Prevent Gastrointestinal Bleeding in Patients With Acute Myocardial Infarction (HELP-MI SWEDEHEART)
Brief Title: HELicobacter Pylori Screening to Prevent Gastrointestinal Bleeding in Patients With Acute Myocardial Infarction
Acronym: HELP-MI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); The Swedish Research Council (Other Government); Hjärt-Lungfonden, Sweden (Unknown)
Responsible Party: Principal Investigator, Robin Hofmann, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: HELP-MI SWEDEHEART
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Infarction; Helicobacter Pylori Infection; GastroIntestinal Bleeding; Cardiovascular Diseases
Keywords: Myocardial infarction; Helicobacter Pylori Infection; GastroIntestinal Bleeding; Cardiovascular Diseases; Registry based randomized clinical trial; Mortality; Cluster-randomized crossover trial
MeSH Terms: conditions — Myocardial Infarction; Gastrointestinal Hemorrhage; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Cluster-randomized, crossover, registry-based clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to randomized cluster assignment of screening/observation period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Helicobacter pylori screening (Active Comparator): At centers randomized to screening, all patients with confirmed MI will be offered H. pylori screening with a bedside UBT incorporated into MI routine care during the hospitalization period. All H. pylori analysis equipment will be supplied by the study organizers, and all centers will use the same equipment (Kibion® Diabact®, Mayoly Spindler, Chatou, France). For patients testing H. pylori positive, eradication therapy will be prescribed at the caring physician's discretion. Control of successful H. pylori eradication therapy with either UBT or H. pylori-antigen in feces 6 weeks after completed eradication therapy will be recommended to the treating physician but not centrally followed-up. The individual implementation of H. pylori screening, test result and eradication therapy prescription will be recorded in SWEDEHEART.
  Interventions: Diagnostic Test: Urea breath test (UBT)
- Usual care without Helicobacter pylori screening (No Intervention): At centers randomized to no screening, all MI patients will receive usual care and will be followed in SWEDEHEART and national registries.

INTERVENTIONS:
Diagnostic Test: Urea breath test (UBT) — After fasting for six hours prior to testing, the patient swallows a C13 Urea tablet or solution and waits. After 10 minutes, the patient exhales and breath is collected (breath bag). The production of 13CO2 is measured by a desktop analyzer (infrared mass spectrometry) and active H. pylori infection diagnosis is made based on previously established cut-off levels for H. pylori infection.
  In patients tested positive, eradication therapy according to the national society of gastroenterology guidelines will be prescribed at the caring physician's discretion.
  Control of successful H. pylori eradication 6 weeks after completed eradication therapy is recommended to the treating physician.
  During the period without H. pylori screening, the study´s UBT equipment will not be available.
  Arms: Helicobacter pylori screening

SUMMARY:
Background: Potent antithrombotic therapy has improved prognosis for patients with acute myocardial infarction (MI) significantly, however, at a price of increased bleeding risk. Helicobacter pylori (H. pylori) infection commonly causes upper gastrointestinal bleeding (UGIB). If systematic screening for H. pylori significantly reduces the risk of UGIB and improves outcomes is unknown.

Study design: A cluster randomized, cross-over, registry-based clinical trial using nationwide Swedish registries for study population definition and data collection.

Population: Patients discharged alive after hospitalization for acute type 1 MI at up to 40 hospitals across Sweden.

Regional PCI networks comprise 18 clusters. Clusters will be randomized to routine H. pylori screening or no screening for 1 year after which cross-over to the opposite strategy occurs for 1 year. The study ends after one additional year of registry-based follow-up, one year after the end of the second period.

Intervention: All MI patients will routinely be offered screening for H. pylori by urea breath test.

Controls: Standard clinical practice. Data will be collected from SWEDEHEART and national registries.

For patients testing H. pylori positive, eradication therapy will be prescribed at the caring physician's discretion. The individual implementation of H. pylori screening, test result and eradication therapy prescription will be recorded in SWEDEHEART. All follow-up data is collected from SWEDEHEART and national registries.

Outcome: Primary outcome is UGIB defined as hospitalization or an outpatient visit in specialized care with ICD codes corresponding to UGIB.

The secondary endpoints (in hierarchical) order:

1. Net Adverse Clinical Events (NACE): All-cause death, UGIB, hospitalization for MI, or hospitalization for ischemic stroke.
2. Major Adverse Cardiovascular and Cerebrovascular Events (MACCE): CV death, hospitalization for MI, or hospitalization for ischemic stroke.
3. All-cause death.
4. CV death.
5. Hospitalization for MI.
6. Hospitalization for stroke.
7. Hospitalization for HF.
8. UGIB requiring blood transfusion.

DETAILED DESCRIPTION:
Background:

Despite progressively reduced mortality over the last decades, cardiovascular disease remains the most common cause of death in both men and women in Sweden and the world. Ischemic heart disease with its acute presentation myocardial infarction (MI) accounts for the majority of cases, approximately 25000 hospitalized patients in Sweden annually.

In addition to early revascularization therapy, potent antithrombotic therapy is the basis for the reduction in cardiovascular events, however, at a price of increased risk of bleeding, typically upper gastrointestinal bleeding (UGIB) that result in substantial morbidity, mortality, and medical care cost. Consequently, antithrombotic therapy may be interrupted in these cases leading to an excessive risk of cardiovascular events; in particular in patients with high age or comorbidities who - by fear of bleeding - rarely receive full recommended treatment from the start. It is recognized that major bleeding events affect prognosis comparably to spontaneous ischemic complications.

To optimize the sensitive trade-off between ischemia and bleeding, risk factor management is crucial. On top of established risk factors - high age, male sex, smoking, dyslipidemia, hypertension, hyperglycemia, physical inactivity - active infection with Helicobacter pylori (H. pylori) may be important for two reasons: First, as it commonly causes acute and chronic gastroduodenal lesions, concomitant anticoagulation or antithrombotic therapy aggravates the risk for bleeding, 2-fold with low dose aspirin, and 7-fold with dual antiplatelet therapy, which today is standard treatment for 12 months post MI. Non-invasive screening for H. pylori can be performed easily by urea breath test (UBT). If found positive, eradication by triple therapy is well established, recommended in risk individuals and believed to reverse the bleeding risk almost completely. Second, H. pylori has been proposed as a causal factor between atherosclerosis progression and plaque instability associated with a two-fold increased risk.

H. pylori may hence be an overlooked risk factor for bleeding complications in MI patients, which potentially could be controlled by routine H. pylori screening. This would be anticipated not only to reduce the UGIB complications after MI but also to improve the adherence to dual antiplatelet therapy and consequently potentially also improve the cardiovascular prognosis in this group.

In summary, the utility of routine H. pylori screening in a contemporary MI population remains undetermined as it is unknown if systematic H. pylori screening reduces the risk of bleeding and improves prognosis.

OBJECTIVE - paradigm and main hypothesis The aim is to determine whether systematic screening for H. pylori after acute MI significantly reduces the risk of UGIB, cardiovascular events and mortality.

STUDY POPULATIONS:

1. PRIMARY INTENTION-TO-TREAT (ITT) POPULATION All adult patients (>18 years of age) registered in SWEDEHEART as discharged alive at a study site with a diagnosis of type 1 MI (including ICD-10 code I21 or I22) analyzed according to randomization.
2. SECONDARY PER-POPULATION (PP) analyses All adult patients (>18 years of age) registered in SWEDEHEART as discharged alive at a study site with a diagnosis of type 1 MI (including ICD-10 code I21 or I22) who were screened for H. pylori (including subcategories screened y/n; screened positive y/n; eradicated y/n if screened positive) are compared to a latent population in the control group from study sites randomized to no-screening.

OUTCOMES All clusters will be analyzed as randomized, irrespective of whether individual patients underwent screening, in accordance with ITT principle. All endpoints in HELP-MI SWEDEHEART are listed below.

The primary endpoint is UGIB defined by appearance of ICD codes obtained from the mandatory National Patient Registry. No central adjudication of events will be performed.

Secondary endpoints are all-cause and cardiovascular mortality, rehospitalization with MI, hospitalization with stroke or heart failure.

MI during the initial hospital stay and readmission due to a nonfatal MI during the first month, will be collected from SWEDEHEART. After day 31, rehospitalization for MI will be captured in the National Patient Registry. All-cause death will be obtained from the Swedish population registry.

Cardiovascular death will be obtained from the Cause-of-death registry. Hospitalization for heart failure and stroke will be obtained from the National Patient Registry.

Tertiary endpoints in patients <80 years of age participating in the routine SWEDEHEART post MI follow-up include symptoms (CCS, NYHA), health related quality of life (EQ5-D index, EQ-VAS, individuals components of EQ-5D), and change in blood glucose (plasma glucose, HbA1c) and blood lipids (total cholesterol, HDL, LDL, triglycerides) from baseline levels at index hospitalization to 6-10 weeks and 11-13 months follow-up.

Health economics based on cost-effectiveness analysis will be performed after one year and including long-term modelling.

The linkage with the National Patient Registry, the National Cause of Death Registry, National Prescribed Drug Registry (prescribed and dispensed treatments), and Statistics Sweden (socioeconomic data) will be done at the end of follow-up.

Pre-specified subgroups are:

* Age
* Sex
* Smoking status
* Hypertension
* Diabetes
* Previous atherosclerotic cardiovascular disease (MI, stroke, peripheral arterial disease)
* Anemia (previous diagnosis and at arrival during index hospitalization)
* Previous gastroduodenal disease (UGIB, peptic ulcer disease, atrophic gastritis, mucosa-associated lymphoid tissue lymphoma, gastric cancer)
* Previous cancer (excluding non-melanoma skin cancer)
* Previous alcohol use disorder
* Chronic or current kidney disease
* MI patients by subcategory (STEMI; NSTEMI)
* MI patients according to revascularization status
* MI patients according to revascularization technique
* Degree of coronary artery disease
* Inflammation (CRP)
* Concomitant medication (antithrombotic, anticoagulation, NSAID, serotonin reuptake inhibitors, cortisone, proton pump inhibitors)
* Planned time on DAPT
* Bleeding risk (using PRECISE DAPT)
* Trial cluster
* Socioeconomic and sociodemographic parameters (region of birth, education level, income)

STATISTICS:

All enrolled patients discharged alive will be included in the primary ITT analyses. Secondary per-protocol analyses will be performed.

The primary analysis is a cluster-summary analysis. In a secondary sensitivity analysis, the outcome will be analyzed using Cox proportional hazards models. The primary analysis (cluster-summary using all follow-up time) of the primary and secondary endpoints will be adjusted for multiplicity using a hierarchical strategy, ordering the endpoints as indicated below.

Prespecified subgroup analysis to determine heterogeneity of treatment effect will be performed but not all included in the primary report.

The primary analysis will use all available follow-up time, censoring patients 2025-01-17. This corresponds to a maximum follow-up time of 3 years + 2 months.

In a sensitivity analysis, follow-up will begin on the admission date rather than the discharge date. Patients who die during hospitalization will not be excluded.

In a set of supplementary analyses, patients will be censored as follows:

* After 30 days.
* After 1 year.
* Censor patients 1 year after the end of the inclusion time for their respective period (Period 1 or 2).
* A landmark analysis, starting the follow-up 30 days after discharge, excluding patients with an event during these 30 days.

All described endpoints will also be analyzed in all subgroups and study populations and reported as above at a later stage. Moreover, long-term (5 years, 10 years) follow-up is planned subsequently.

A detailed statistical analysis plan with prespecified analyses will be published alongside the primary report.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Registered in SWEDEHEART as discharged alive at a study site with a diagnosis of type 1 MI (including ICD-10 code I21 or I22).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2030-01-17 (Estimated)

PRIMARY OUTCOMES:
Upper gastrointestinal bleeding (UGIB) | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to UGIB

SECONDARY OUTCOMES:
Net Adverse Clinical Events (NACE) | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to all-cause death, UGIB, hospitalization with MI, or hospitalization for ischemic stroke (NACE).
Major Adverse Cardiac or Cerebrovascular Events (MACCE) | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to cardiovascular death, rehospitalization with MI, or hospitalization for ischemic stroke (MACCE)
All-cause death | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to all-cause death
Cardiovascular death | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to cardiovascular death
Rehospitalization with myocardial infarction | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to rehospitalization with myocardial infarction
Hospitalization for ischermic stroke | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to hospitalization for ischemic stroke
Hospitalization for heart failure | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to hospitalization for heart failure
UGIB requiring blood transfusion | Time from discharge date of index MI hospitalization to the end of study follow-up, January 17, 2025 (corresponds to a maximum follow-up time of 3 years and 2 months, and minimum of 1 year).
  Time from discharge date of index MI hospitalization to UGIB requiring blood transfusion

OTHER OUTCOMES:
CCS | 6-10 weeks after discharge date of index MI hospitalization
  Symptoms of angina and functional status (CCS class) at 6-10 weeks after discharge date of index MI hospitalization
CCS | 11-13 months after discharge date of index MI hospitalization
  Symptoms of angina and functional status (CCS class) at 11-13 months after discharge date of index MI hospitalization
NYHA | 6-10 weeks after discharge date of index MI hospitalization
  Symptoms of dyspnea and functional status (NYHA class) at 6-10 weeks after discharge date of index MI hospitalization
NYHA | 11-13 months after discharge date of index MI hospitalization
  Symptoms of dyspnea and functional status (NYHA class) at 11-13 months after discharge date of index MI hospitalization
Blood lipids | Change from baseline levels during index hospitalization to 6-10 weeks after discharge date of index MI hospitalization
  Total cholesterol, HDL, LDL and triglycerides (mmol/L) at 6-10 weeks after discharge date of index MI hospitalization.
Blood lipids | Change from baseline levels during index hospitalization to 11-13 months after discharge date of index MI hospitalization
  Total cholesterol, HDL, LDL and triglycerides (mmol/L) at 11-13 months after discharge date of index MI hospitalization.
Plasma glucose | Change from baseline levels during index hospitalization to 6-10 weeks after discharge date of index MI hospitalization
  Plasma glucose (mmol/L) at 6-10 weeks after discharge date of index MI hospitalization.
Plasma glucose | Change from baseline levels during index hospitalization to 11-13 months after discharge date of index MI hospitalization
  Plasma glucose (mmol/L) at 11-13 months after discharge date of index MI hospitalization.
Hb1Ac | Change from baseline levels during index hospitalization to 6-10 weeks after discharge date of index MI hospitalization
  Hb1Ac (mmol/mol) at 6-10 weeks after discharge date of index MI hospitalization.
Hb1Ac | Change from baseline levels during index hospitalization to at 11-13 months after discharge date of index MI hospitalization
  Hb1Ac (mmol/mol) at at 11-13 months after discharge date of index MI hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Hofmann, MD, PhD, Principal Investigator — Karolinska Institutet, Department of Clinical Science and Education, Södersjukhuset, Stockholm.
Locations (35):
- Sweden (35):
  - Södra Älvsborg Hospital, Borås
  - Eskilstuna Hospital, Eskilstuna
  - Falun Hospital, Falun
  - Gävle Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Östra Hospital, Gothenburg
  - Halmstad Hospital, Halmstad
  - Helsingborg Hospital, Helsingborg
  - Ryhov Hospital, Jönköping
  - Karlskrona Hospital, Karlskrona
  - Köping Hospital, Köping
  - Kristianstad Hospital, Kristianstad
  - Kungälv Hospital, Kungälv
  - Lidköping Hospital, Lidköping
  - Linköping University Hospital, Linköping
  - Skåne University Hospital Lund, Lund
  - Skåne University Hospital Malmö, Malmo
  - Mora Hospital, Mora
  - Motala Hospital, Motala
  - Mölndal Hospital, Mölndal
  - Vrinnevisjukhuset, Norrköping
  - Norrtälje Hospital, Norrtälje
  - Nyköping Hospital, Nyköping
  - Örebro University Hospital, Örebro
  - Sunderby Hospital, Södra Sunderbyn
  - Danderyds University Hospital, Stockholm
  - Karolinska University Hospital Huddinge, Stockholm
  - Karolinska University Hospital Solna, Stockholm
  - Sankt Görans Hospital, Stockholm
  - Södersjukhuset, Stockholm
  - Norra Älvsborgs Länssjukhus, Trollhättan
  - Norrland University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
  - Varberg Hospital, Varberg
  - Västerås Hospital, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofmann R, Back M. Time for Routine Helicobacter pylori Screening in Coronary Artery Disease? Circulation. 2023 Jun 6;147(23):1731-1733. doi: 10.1161/CIRCULATIONAHA.123.064944. Epub 2023 Jun 5. No abstract available. PMID 37276250
- [Background] Sundqvist MO, Warme J, Hofmann R, Pawelzik SC, Back M. Helicobacter Pylori Virulence Factor Cytotoxin-Associated Gene A (CagA) Induces Vascular Calcification in Coronary Artery Smooth Muscle Cells. Int J Mol Sci. 2023 Mar 11;24(6):5392. doi: 10.3390/ijms24065392. PMID 36982467
- [Background] Warme J, Sundqvist MO, James S, Hofmann R. Screening for Helicobacter pylori infection in patients with cardiovascular and gastrointestinal disease. Nat Rev Cardiol. 2024 Aug;21(8):593. doi: 10.1038/s41569-024-01028-8. No abstract available. PMID 38698181
- [Background] Capodanno D, Bhatt DL, Gibson CM, James S, Kimura T, Mehran R, Rao SV, Steg PG, Urban P, Valgimigli M, Windecker S, Angiolillo DJ. Bleeding avoidance strategies in percutaneous coronary intervention. Nat Rev Cardiol. 2022 Feb;19(2):117-132. doi: 10.1038/s41569-021-00598-1. Epub 2021 Aug 23. PMID 34426673
- [Background] Lanas A, Santilli F. Aspirin and Helicobacter pylori interaction. Lancet. 2022 Nov 5;400(10363):1560-1561. doi: 10.1016/S0140-6736(22)02000-1. No abstract available. PMID 36335960
- [Background] Hawkey C, Avery A, Coupland CAC, Crooks C, Dumbleton J, Hobbs FDR, Kendrick D, Moore M, Morris C, Rubin G, Smith M, Stevenson D; HEAT Trialists. Helicobacter pylori eradication for primary prevention of peptic ulcer bleeding in older patients prescribed aspirin in primary care (HEAT): a randomised, double-blind, placebo-controlled trial. Lancet. 2022 Nov 5;400(10363):1597-1606. doi: 10.1016/S0140-6736(22)01843-8. PMID 36335970
- [Background] Mascellino MT, Pontone S, Vega AE, Malfertheiner P. Editorial: Helicobacter pylori infection: pathogenesis, antibiotic resistance, advances and therapy, new treatment strategies. Front Microbiol. 2022 Dec 8;13:1102144. doi: 10.3389/fmicb.2022.1102144. eCollection 2022. No abstract available. PMID 36569072
- [Background] Malfertheiner P, Megraud F, Rokkas T, Gisbert JP, Liou JM, Schulz C, Gasbarrini A, Hunt RH, Leja M, O'Morain C, Rugge M, Suerbaum S, Tilg H, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study group. Management of Helicobacter pylori infection: the Maastricht VI/Florence consensus report. Gut. 2022 Aug 8:gutjnl-2022-327745. doi: 10.1136/gutjnl-2022-327745. Online ahead of print. PMID 35944925
- [Background] Talasaz AH, Sadeghipour P, Ortega-Paz L, Kakavand H, Aghakouchakzadeh M, Beavers C, Fanikos J, Eikelboom JW, Siegal DM, Monreal M, Jimenez D, Vaduganathan M, Castellucci LA, Cuker A, Barnes GD, Connors JM, Secemsky EA, Van Tassell BW, De Caterina R, Kurlander JE, Aminian A, Piazza G, Goldhaber SZ, Moores L, Middeldorp S, Kirtane AJ, Elkind MSV, Angiolillo DJ, Konstantinides S, Lip GYH, Stone GW, Cushman M, Krumholz HM, Mehran R, Bhatt DL, Bikdeli B. Optimizing antithrombotic therapy in patients with coexisting cardiovascular and gastrointestinal disease. Nat Rev Cardiol. 2024 Aug;21(8):574-592. doi: 10.1038/s41569-024-01003-3. Epub 2024 Mar 20. PMID 38509244
- [Background] Sarri GL, Grigg SE, Yeomans ND. Helicobacter pylori and low-dose aspirin ulcer risk: A meta-analysis. J Gastroenterol Hepatol. 2019 Mar;34(3):517-525. doi: 10.1111/jgh.14539. Epub 2018 Dec 17. PMID 30408229
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Lindholm D, Sarno G, Erlinge D, Svennblad B, Hasvold LP, Janzon M, Jernberg T, James SK. Combined association of key risk factors on ischaemic outcomes and bleeding in patients with myocardial infarction. Heart. 2019 Aug;105(15):1175-1181. doi: 10.1136/heartjnl-2018-314590. Epub 2019 May 4. PMID 31055499
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Shestakovska O, Aboyans V, Alings M, Anand SS, Avezum A, Berkowitz SD, Bhatt DL, Cook-Bruns N, Felix C, Fox KAA, Hart RG, Maggioni AP, Moayyedi P, O'Donnell M, Ryden L, Verhamme P, Widimsky P, Zhu J, Yusuf S. Bleeding and New Cancer Diagnosis in Patients With Atherosclerosis. Circulation. 2019 Oct 29;140(18):1451-1459. doi: 10.1161/CIRCULATIONAHA.119.041949. Epub 2019 Sep 12. PMID 31510769
- [Background] Fang Y, Fan C, Xie H. Effect of Helicobacter pylori infection on the risk of acute coronary syndrome: A systematic review and meta-analysis. Medicine (Baltimore). 2019 Dec;98(50):e18348. doi: 10.1097/MD.0000000000018348. PMID 31852134
- [Background] Ng JC, Yeomans ND. <em>Helicobacter pylori</em> infection and the risk of upper gastrointestinal bleeding in low dose aspirin users: systematic review and meta-analysis. Med J Aust. 2018 Sep 1;209(7):306-311. doi: 10.5694/mja17.01274. PMID 30257623
- [Background] Chey WD, Leontiadis GI, Howden CW, Moss SF. ACG Clinical Guideline: Treatment of Helicobacter pylori Infection. Am J Gastroenterol. 2017 Feb;112(2):212-239. doi: 10.1038/ajg.2016.563. Epub 2017 Jan 10. PMID 28071659
- [Background] Xu Z, Li J, Wang H, Xu G. Helicobacter pylori infection and atherosclerosis: is there a causal relationship? Eur J Clin Microbiol Infect Dis. 2017 Dec;36(12):2293-2301. doi: 10.1007/s10096-017-3054-0. Epub 2017 Jul 27. PMID 28752210
- [Background] Warme J, Sundqvist M, Mars K, Aladellie L, Pawelzik SC, Erlinge D, Jernberg T, James S, Hofmann R, Back M. Helicobacter pylori screening in clinical routine during hospitalization for acute myocardial infarction. Am Heart J. 2021 Jan;231:105-109. doi: 10.1016/j.ahj.2020.10.072. Epub 2020 Nov 2. PMID 33144087
- [Background] Hellstrom PM, Benno P, Malfertheiner P. Gastrointestinal bleeding in patients with Helicobacter pylori and dual platelet inhibition after myocardial infarction. Lancet Gastroenterol Hepatol. 2021 Sep;6(9):684-685. doi: 10.1016/S2468-1253(21)00192-8. No abstract available. PMID 34391514
- [Background] Sarajlic P, Simonsson M, Jernberg T, Back M, Hofmann R. Incidence, associated outcomes, and predictors of upper gastrointestinal bleeding following acute myocardial infarction: a SWEDEHEART-based nationwide cohort study. Eur Heart J Cardiovasc Pharmacother. 2022 Aug 11;8(5):483-491. doi: 10.1093/ehjcvp/pvab059. PMID 34423350
- [Derived] Hofmann R, James S, Sundqvist MO, Warme J, Angeras O, Alfredsson J, Erlinge D, Arefalk G, Arstad G, Blomberg S, Frobert O, Hambraeus K, Hellstrom PM, Lauermann J, Lidin M, Lindhagen L, Mourtzinis G, Schoede C, Thunstrom E, Voldberg B, Wagner H, Ostlund O, Jernberg T, Back M. Helicobacter pylori Screening After Acute Myocardial Infarction: The Cluster Randomized Crossover HELP-MI SWEDEHEART Trial. JAMA. 2025 Oct 7;334(13):1160-1169. doi: 10.1001/jama.2025.15047. PMID 40887995
- [Derived] Hofmann R, James S, Sundqvist MO, Warme J, Frobert O, Angeras O, Hellstrom PM, Hambraeus K, Alfredsson J, Erlinge D, Lauermann J, Lindhagen L, Ostlund O, Jernberg T, Back M. HELicobacter Pylori screening to prevent gastrointestinal bleeding in patients with acute Myocardial Infarction (HELP-MI SWEDEHEART) - Design and rationale of a cluster randomized, crossover, registry-based clinical trial. Am Heart J. 2025 Aug;286:66-74. doi: 10.1016/j.ahj.2025.03.014. Epub 2025 Mar 27. PMID 40157409